CLINICAL TRIAL: NCT04914923
Title: Mindfulness-Based Interventions for OCD: Efficacy, Mechanisms, and Biological Predictors of Outcome
Brief Title: Mindfulness-Based Interventions for OCD
Acronym: MindOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other); McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RN440237-452052
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Cognitive Behaviour Therapy; Mindfulness-based Intervention; Mindfulness-based cognitive therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy; Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: Treatment-seeking participants at Sunnybrook Health Sciences Centre (SHSC) and St. Joseph's Healthcare Hamilton, McMaster University (McMaster) with a primary DSM-5 diagnosis of OCD will be randomly assigned to receive a: 1) 12-week MBCT group intervention, 2) a 12-week CBT intervention or 3) a 12-week waitlist condition and will complete repeated assessments at baseline, throughout treatment, at post-treatment and three-month follow-up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive Behaviour Therapy (Experimental): This study arm will receive 12 weeks of cognitive behaviour therapy as an intervention.
  Interventions: Behavioral: Cognitive Behaviour Therapy (CBT)
- Mindfulness-based Cognitive Therapy (Experimental): This study arm will receive 12 weeks of a mindfulness-based cognitive therapy intervention, along with open mindfulness sessions via an EEG headset.
  Interventions: Device: Muse; Behavioral: Mindfulness-Based Cognitive Therapy (MBCT)
- Waitlist (No Intervention): This study arm will not receive an intervention for 12 weeks.

INTERVENTIONS:
Device: Muse — Muse is an EEG headset device created by Interaxxon to track brain waves during mindfulness sessions.
  Arms: Mindfulness-based Cognitive Therapy
Behavioral: Cognitive Behaviour Therapy (CBT) — Cognitive behavioural therapy (CBT), incorporating exposure/response prevention (ERP) and cognitive therapy, is considered the gold-standard treatment for OCD. The efficacy of CBT has been well established, with numerous studies demonstrating that it leads to significant and lasting reduction in OCD symptoms for the majority of completers.
  Arms: Cognitive Behaviour Therapy
Behavioral: Mindfulness-Based Cognitive Therapy (MBCT) — Mindfulness-based interventions (MBIs) including MBCT, are interventions that incorporate formal and informal mindfulness practice in order to treat mental health concerns.
  Arms: Mindfulness-based Cognitive Therapy

SUMMARY:
Obsessive-compulsive disorder (OCD) is a severe and debilitating anxiety disorder afflicting about 2% of the population. It is characterized by the presence of recurrent obsessions and/or compulsions that are time consuming and cause marked distress and/or impairment. Untreated, OCD runs a chronic and deteriorating course. According to the World Health Organization, OCD is among the top 10 leading causes of disability worldwide. Examination of non-medicinal treatments for OCD has focused on two distinct treatments: exposure and response prevention (ERP) and cognitive therapy (CT), often combined into an integrated cognitive-behavioural treatment (CBT). CBT is considered the first line psychological treatment for OCD, with estimates of response rates of between 70-80%. However, there are a significant number of treatment non-responders and the majority of responders are still left with impairing residual symptoms. One area of investigation that has shown potential benefit for general mood and anxiety disorders has been mindfulness-based interventions (MBIs), yet the potential benefits of MBIs in OCD has been largely unexamined, except for several small preliminary studies that show clinical promise. The purpose of this study is to examine the clinical benefits of a standardized MBI treatment for OCD in a large-scale, multi-site randomized controlled trial. The results of this study will directly determine whether Mindfulness can be considered an effective treatment for OCD. If this study can demonstrate that a short-term mindfulness intervention can significantly reduce the suffering associated with OCD, then the findings could easily be translated into routine clinical care in and out of hospital settings. Results of this study will also potentially add to our understanding of the mechanisms that drive OCD symptoms, improve our knowledge of psychological treatment mechanisms, and elucidate how biological factors influence psychological treatment outcomes.

DETAILED DESCRIPTION:
Cognitive Behavioural Therapy (CBT) is a first line psychological treatment for OCD with estimated response rates of between 70-80%. However, there are still a substantial number of treatment non-responders and the vast majority of responders are left with impairing residual symptoms. One new area of investigation that has shown potential benefit for the treatment of OCD has been mindfulness-based interventions (MBIs). This emerging literature provides proof of principle for the delivery and potential efficacy of MBIs for OCD, particularly as an adjunct to CBT, with all studies reporting large (d > .80) treatment effects. To date, only our teams' small, non-controlled pilot study (N=19) has shown promise for a MBI as a stand-alone treatment for OCD separate from CBT (d = 1.10). However, all results to date for MBI treatments for OCD must be interpreted with caution as they have utilized small, underpowered sample sizes, have not included control groups, and failed to control for potentially confounding variables (e.g., medications, self-initiated exposures). The proposed four-year, two-site randomized controlled trial at two of Canada's leading OCD treatment centres (Sunnybrook Health Sciences Centre and St. Joseph's Healthcare Hamilton) that have been involved in developing and piloting MBI treatments for OCD will aim to test whether a structured, Mindfulness-Based Cognitive Therapy (MBCT) intervention for OCD is an efficacious treatment for a large, heterogeneous sample of DSM-5 (Diagnostic Statistical Manual of Mental Disorders 5th edition) diagnosed OCD participants. The primary aim of this proposed study is to examine whether a developed and piloted MBCT treatment for OCD is efficacious when compared to a waitlist condition and to explore its efficacy compared to CBT treatment for OCD. A secondary aim of the study is to examine the putative treatment mechanisms of MBCT. Past research examining treatment mechanisms in CBT for OCD have focused on the reduction of obsessional beliefs, anxiety sensitivity, and safety behaviours in producing better outcomes. In contrast, the hypothesized mechanisms in MBI treatments include the development of mindfulness skills such as acting with awareness, non-reactivity to and non-judging of inner experience, and reduction in mind wandering. The large-scale, powered RCT (randomized control trial) design will permit the examination of whether MBCT and CBT include overlapping or distinct treatment mechanisms. Treatment outcomes will be assessed with standardized measures of OCD symptomatology, general measures of mood and anxiety, a reliable and valid EEG measure to assess cognitive changes across treatment. If this study can demonstrate that a short-term mindfulness intervention can significantly reduce the suffering associated with OCD, then the findings could easily be translated into routine clinical care in and out of Canadian hospital settings. Results of this study will also potentially add to our understanding of the mechanisms that drive OCD symptoms, improve our knowledge of psychological treatment mechanisms, and elucidate how genetic/biological factors influence psychological treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* experiencing clinically significant obsessive-compulsive symptoms based on the Yale-Brown Obsessive Compulsive Scale (YBOCS; score > 17)
* if on medications for OCD, must be stabilized, i.e. are currently receiving an adequate dose (equivalent of 40mg/day of fluoxetine) for an adequate duration (at least 8 weeks of treatment) prior to the initiation of the study.

Exclusion Criteria:

* concurrent diagnosis of a severe mood disorder, schizophrenia or other psychotic disorders, or substance abuse/dependence
* suspected organic pathology
* an active comorbid medical condition that may require urgent intervention during the treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in OCD symptom severity, as measured by the Yale-Brown Obsessive Compulsive Scale (YBOCS) | Baseline to 12 weeks
  OCD symptom severity will be measured using the Yale-Brown Obsessive Compulsive Scale (YBOCS).The YBOCS is a standardized rating scale measuring 10 items pertaining to obsessions and compulsions on a 5-point Likert scale ranging from 0 (no symptoms) to 4 (severe symptoms). Both the self-report and clinician interview versions of the YBOCS have been shown to possess high internal consistency and validity.

SECONDARY OUTCOMES:
Change from baseline in OCD symptomatology, as measured by the OCI-R (Obsessive Compulsive Inventory - Revised). | Baseline to 12 weeks
  This self -report short version of the OCI consisting of 18 items measures six distinct factors: Washing, Checking, Ordering, Obsessing, Hoarding and Neutralizing, to chart the change in OCD symptomatology across time.
Change from baseline in the experience of depression, anxiety and stress symptoms, as measured by the DASS-21 (Depression, Anxiety and Stress Scale - 21 items). | Baseline to 12 weeks
  Depression, anxiety and stress severity will be measured using the Depression Anxiety Stress Scales-21,a self-report questionnaire comprising three subscales with seven items each for depression, anxiety and stress. The DASS-21 shows high internal consistency, high reliability in distinguishing between depression, anxiety and stress in adults, and good convergent and discriminant validity.
Change from baseline in various attitudes and beliefs related to obsessional thoughts, as measured by the OBQ-44 (Obsessional Beliefs Questionnaire - 44 items). | Baseline to 12 weeks
  The Obsessional Beliefs Questionnaire is a 44-item self-report questionnaire designed to assess the extent to which respondents agree or disagree with various attitudes and beliefs related to obsessional thoughts. The OBQ is internally consistent, and evidences good test-retest reliability, convergent validity, and discriminant validity.
Change from baseline in aspects of mindfulness, as measured by the FFMQ (Five Facet Mindfulness Questionnaire). | Baseline to 12 weeks
  The Five Facet Mindfulness Questionnaire is a self-report questionnaire containing 39 items that assess five aspects of mindfulness: observing, describing, acting with awareness, non-judgment of inner experiences, and non-reactivity to inner experience.
Change from baseline in functional health and well-being, as measured by the SF-36 Health Survey (Short Form 36 item Health Survey). | Baseline to 12 weeks
  The SF-36 Health Survey is a brief questionnaire containing 36 items about functional health and well-being. The reliability and validity of the SF-36 have been well documented. It has demonstrated good treatment sensitivity
Change from baseline in the degree which individuals find distress intolerable, as measured by the DTS (Distress Tolerance Scale). | Baseline to 12 weeks
  The Distress Tolerance Scale is a 15-item self-report questionnaire that measures the degree to which individuals find distress intolerable, unacceptable, impairing, and necessary to avoid. Distress tolerance has been linked to OCD.
Change from baseline in the fear of consequences of anxiety, as measured by the ASI-3 (Anxiety Sensitivity Index). | Baseline to 12 weeks
  The Anxiety Sensitivity Index-3 is an 18-item self-report measure of the degree to which individuals fear the consequences of anxiety. It is composed of three subscales: fear of the physical, social, and cognitive consequences of anxiety.
Change from baseline in the time spent ruminating, as measured by the RRS (Ruminative Response Scale). | Baseline to 12 weeks
  The Ruminative Response Scale is a frequently used 22-item measure of the amount to which participants are engaging in rumination, or repetitive, passive, and negative self-focus.

OTHER OUTCOMES:
Change from baseline in OCD symptomatology, as measured by the EEG headset device "Muse". | Baseline to 12 weeks
  Participants will be instructed to use the "Muse" EEG headset for open, unguided mindfulness sessions. The device will measure alpha and beta band oscillatory power and how it will change over the 12 weeks of treatment intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Rector, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No